CLINICAL TRIAL: NCT03409952
Title: Evaluation of the Lutronic LaseMD System for the Treatment of Benign Pigmented Lesions
Brief Title: Lutronic LaseMD for Treatment of Benign Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: L17001
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Benign Pigmented Lesions
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled first into Group A, then Group B will be enrolled. Subjects may not be enrolled in both groups.
Who Masked: Outcomes Assessor
Masking Description: Group A: Three blinded physician evaluators will assess an identical set of split side post-treatment photos, comparing the left and right photo for improvement in benign pigmented lesions.
  Group B: Three blinded physician evaluators will assess an identical set of pre-treatment and post-treatment photos, comparing the left and right photo for improvement in benign pigmented lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: LaseMD and DUAL 1927nm Laser (Active Comparator): Group A subjects will receive split-side study treatments comparing two devices: LaseMD compared to the DUAL 1927nm laser.
  Interventions: Device: LaseMD and DUAL 1927nm Laser
- Group B: LaseMD Optimized (Active Comparator): Group B subjects will receive LaseMD Optimized Treatments based on Group A treatment data.
  Interventions: Device: LaseMD

INTERVENTIONS:
Device: LaseMD and DUAL 1927nm Laser — Laser treatment of benign pigmented lesion based on photothermolysis whereby the target molecule, the chromophore, absorbs a delivered wavelength of light over a period of time to damage the target while limiting collateral damage to adjacent structures, leading to pigmentary clearance.
  Arms: Group A: LaseMD and DUAL 1927nm Laser
Device: LaseMD — Laser treatment of benign pigmented lesion using optimized treatment settings.
  Arms: Group B: LaseMD Optimized

SUMMARY:
The Lutronic LaseMD Laser System will be evaluated for the treatment of benign pigmented lesions.

DETAILED DESCRIPTION:
This clinical trial is a designed as a prospective, multi-site, non-randomized study of 20 subjects and two treatment groups. Subjects will be enrolled first into Group A, then Group B.

Group A: LaseMD 100 Tip Random Mode vs. DUAL 1927nm (n=12) Group A subjects will receive a split treatment of the décolleté, with LaseMD treatment on one side and DUAL 1927 treatment on the other side. Post-treatment follow-up visits (Days 4, 7, 14, 28, 90) will be conducted to assess adverse events, expected treatment effects, capture digital images, and assess efficacy.

Group B: LaseMD Optimized Treatments (n=8) Based on safety and efficacy data captured from Group A, subjects in Group B will be treated with the LaseMD optimized treatment parameters for benign pigmented lesions on décolleté, arms, hands, face, and/or neck. A phone follow-up will occur at Day 4 for the assessment of adverse events and expected treatment effects. Post-treatment follow-up visits (Days 4, 7, 14, 28, 90) will be conducted to assess adverse events, expected treatment effects, capture digital images, and assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years and older.
2. Subject in good health.
3. Fitzpatrick Skin Type I to VI.
4. Presence of benign pigmented lesions on décolleté, arms, hands, face, and/or neck.
5. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
6. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
7. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   1. Postmenopausal for at least 12 months prior to study;
   2. Without a uterus and/or both ovaries; or
   3. Bilateral tubal ligation at least six months prior to study enrollment.
8. Absence of physical or psychological conditions unacceptable to the investigator.
9. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
10. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active systemic or local skin disease that may affect wound healing.
2. History of keloids or poor wound healing.
3. Significant scarring in the area(s) to be treated that would interfere with assessing results.
4. Open wounds or lesions in the area(s) to be treated.
5. Inability to understand the protocol or to give informed consent.
6. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within four weeks prior to study participation or during the study.
7. Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
8. History of chronic drug or alcohol abuse.
9. History of collagen vascular disease.
10. History of autoimmune disease.
11. Subjects with implanted pacemaker or defibrillator.
12. Subjects with sensitivity or allergy to gold.
13. Subjects with sensitivity or allergy to benzocaine, lidocaine, ortetracaine.
14. Subjects with photosensitive skin.
15. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
16. Subjects who are pregnant or lactating or anticipate becoming pregnant during the study.
17. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
18. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
19. Concurrent enrollment in any study involving the use of investigational devices or drugs.
20. Current smoker or history of smoking in the last five years.
21. Current user of any nicotine-containing products,e.g.,ecigarettes, Nicorette gum, nicotine patches,etc.
22. History of surgical or cosmetic treatments in the area(s) to be treated within the past 6 months.
23. History or current use of the following prescription medications:

    1. Accutane or other systemic retinoids within the past twelve months;
    2. Topical Retinoids within the past two weeks; and/or
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix).
24. Psychiatric drugs that in the investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Group A: Evaluation of split-side pigmentary clearance | 90 days following the last study treatment
  Blinded assessment of paired post-treatment study photographs conducted by three blinded physician evaluators will compare split-side post-treatment photos. Each assessor will be given identical paired post-treatment photo sets. Each photo's treatment device (LaseMD or DUAL 1927nm) will NOT be marked. Each assessor will compare the Left and Right photo for improvement in benign pigmented lesions using the following definitions:
  Change = an improvement that is striking, substantial and immediately noticeable; readily apparent but modest in nature; or slight and subtle in nature.
  The photo believed to be the most improved photo (Left photo or Right photo) is selected.
Group B: Percentage of pigmentary clearance in standard photographs | 90 days following the last study treatment
  Blinded assessment of paired study photographs conducted by three blinded physician assessors will compare pre- and post-treatment photos. Each assessor will compare paired photo sets for percentage of pigmentary clearance using a score of 0-4: 0=poor (0-24%), 1=fair (25-49%), 2=good (50-74%), 3=excellent (75-95%), 4=complete (95%+) improvement.
  Each assessor will be given identical paired pre- and post-treatment photo sets. Each photo's visit interval (pre and post treatment) will NOT be marked. Each assessor will compare Left and Right photo for improvement in benign pigmented lesions using the following definitions:
  * Change = an improvement that is striking, substantial and immediately noticeable; readily apparent but modest in nature; or slight and subtle in nature.
  The photo believed to be the post-treatment photo (Left photo or Right photo) is selected. The assessor will then score the percentage of pigmentary clearance using the 0-4 scale.

SECONDARY OUTCOMES:
Clinician assessment of overall aesthetic improvement | 28 and 90 days following study treatments
  Overall aesthetic improvement based on completion of the Clinician Global Aesthetic Improvement Scale. Split-side assessments will be conducted for Group A subjects. The scale will be administered based on a live assessment of the subject while referring to the subject's pre-treatment photographs, and based on a comparison of the subject's pre-treatment photographs to the current post-treatment photographs. Aesthetic improvement will be based on the following definitions:
  1. = Improved: Improvement in appearance from initial condition
  2. = No Change: The appearance is essentially the same as the original condition.
  3. = Worse: The appearance is worse than the original condition.
Subject assessment of overall aesthetic improvement | 28 and 90 days following study treatments
  Overall aesthetic improvement based on completion of the Subject Global Aesthetic Improvement Scale. Split-side assessments will be conducted for Group A subjects. Subjects will complete the scale based on a live assessment referring to a hand mirror and their pre-treatment photographs, and based on a comparison of their pre-treatment photographs to the current post-treatment photographs. Aesthetic improvement will be based on the following definitions:
  1. = Improved: Improvement in appearance from initial condition
  2. = No Change: The appearance is essentially the same as the original condition.
  3. = Worse: The appearance is worse than the original condition.
Patient Satisfaction Questionnaire | 90 days following study treatment
  Based on completion of a Patient Satisfaction Questionnaire while referring to a hand mirror and their pre-treatment photographs. Group A subjects will be asked to complete the questionnaire based on a split-side assessment providing responses specific to each treatment side, i.e., LaseMD treated and DUAL 1927mm treated. Patients will be asked to provides responses to document the level of improvement in skin pigment using the following categories of improvement: 75-100% improved, 50-74% improved, 25-49% improved, 0-24% improved; document any other improvements noted, e.g., skin texture improvement, skin tone improvement, fine lines and wrinkles improvement, etc.; characterize their level of satisfaction based on the following levels of satisfaction: Very Satisfied, Satisfied, Slightly Satisfied; Neither Satisfied or Dissatisfied, Dissatisfied; document if they would recommend each treatment to friends and family members.
Treated-related pain | For the duration of each study treatment
  During study treatment, subjects' pain levels will be monitored using a validated Numeric Rating Scale (0-10), with 0 being 'No Pain' and 10 being the 'Worst Possible Pain'. The average pain score for each device will be recorded. Group A will be split-side assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Maryland Dermatology Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - Dermatology, Laser, and Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No